CLINICAL TRIAL: NCT07167186
Title: Evaluation of a Multimodal Day Hospital for the Overall Management of Patients With Chronic Inflammatory Bowel Diseases (IBD)
Acronym: AMBUMIC
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 240469; IDRCB: 2024-A00870-47 (Other: ANSM)
Record Dates: First submitted 2025-06-09; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Disease (IBD); Crohn Disease; Ulcerative Colitis (Disorder)
Keywords: Therapeutic education; Inflammatory bowel disease; Crohn's disease; Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Inflammatory bowel diseases (IBD) are long-term conditions affecting more than 250,000 people in France. They typically begin in young adults and are characterized by flare-ups interspersed with periods of remission. The impact of these diseases goes beyond digestive symptoms, with fatigue present in 50 to 80% of cases. The overall effect on health leads to a decline in quality of life and work productivity. Therapeutic management relies on long-term immunosuppressive treatments aimed at inducing prolonged remission. While therapeutic management has become more complex with an increasing number of available treatments, evaluating the effectiveness and tolerance of these treatments requires a multimodal approach, including therapeutic education and specific follow-up based on the patient's profile and treatment, with the goal of comprehensive care and precision medicine.

Recently, multimodal day hospitalizations have been developed, particularly in response to the recent evolution of treatment administration routes toward subcutaneous or oral forms. In 2022, the gastroenterology and nutrition department of Saint Antoine Hospital, which follows 3,500 patients with CIBD, created a multimodal day hospital (DH) (four interventions) dedicated to patients treated with biologics and Janus kinase inhibitors. In a single session, this approach systematically combines (1) specific biological tests, especially pharmacokinetics, (2) a consultation with a gastroenterologist, (3) a consultation with a therapeutic education nurse, (4) and, depending on the identified needs of the patients, a dietary workshop or fatigue management session; a specialized dermatology or rheumatology consultation; and an ultrasound of the intestinal wall.

The goal of this study is to assess the benefits of a multimodal day hospital on the management and skills of patients with IBD.

DETAILED DESCRIPTION:
This is a non-interventional cohort study. Patients will be included over a 6-month period during a scheduled multimodal day hospital visit as part of their care. Before their day hospital appointment, patients will receive an information sheet explaining the research process.

M0 Inclusion:

Patients who agree to participate in the research will receive evaluation questionnaires to be completed online, which include:

* Access to care,
* Adherence according to the self-declared adherence rate,
* Knowledge about their disease (IBDKID2),
* Fatigue (FACIT-F),
* Dietary questionnaire (SLFQ),
* Productivity (WPAI). Patients who do not wish to participate in the study during their visit to the multimodal day hospital will be excluded from the study.

Day of DH:

Upon arrival at the multimodal day hospital, if the questionnaires have not been completed in advance, patients will be offered the opportunity to complete them during their visit, with an estimated duration of 30 minutes.

M1 (4 Weeks Post-DH):

Four weeks after the day hospital visit, patients will receive an email with a link to complete the questionnaires again (adherence, knowledge of their disease, fatigue, dietary questionnaire, and productivity). If the questionnaires are not completed, a reminder email will be sent 3 days and 1 month after the due date. If there is no response, a phone call will be scheduled 1 week after the initially planned date by the clinical research technician. Questionnaires can be filled out up to 8 weeks after inclusion.

M6 (6 Months Post-DH):

Six months after the day hospital visit, patients will again receive an email with a link to complete the questionnaires (adherence, knowledge of their disease, fatigue, dietary questionnaire, and productivity). A reminder email will be sent 3 days and 1 month after the due date if there is no response. If there is still no response, a phone call will be made 1 week after the initially scheduled date by the clinical research technician. Questionnaires can be completed up to 7 months after inclusion.

Between M0 and M1:

Treatment optimization and the update of the vaccination schedule will be recorded in the patient's electronic health record.

Study Participation End:

Participation in the study will conclude after the completion of the questionnaires, no later than 7 months after inclusion Statistical analysis The analysis will be performed using SAS v9.4 software (or a later version) by the URC-Est at the end of the study after the database freeze. A detailed statistical analysis plan will be written before the database freeze. A flow chart will be created.

The patient profile at inclusion will be described, including comorbidities, characteristics of the IBD (such as clinical and biological activity at the time of the day hospital visit), and treatments. The day hospital process will be evaluated, including the number of patients per session and the type of interventions performed.

Qualitative variables will be described by their frequency and count, while quantitative variables will be described by their mean and standard deviation or by their median and interquartile range, depending on their distribution.

Analysis of the Primary Endpoint The proportion of patients with an improvement in their skills at one month or an improvement in the management of their disease will be calculated. The proportion of patients with improvement in each of the two groups of criteria will also be calculated.

Analysis of Secondary Endpoints Secondary endpoints will be measured by the proportion of patients showing improvement for each individual item. The total number of items with improvement per patient will also be evaluated, as well as the proportion of patients with access to practitioners such as a dietitian specialized in IBD, a rheumatologist, or a dermatologist outside the day hospital, based on the dedicated questionnaire.

A logistic regression will be conducted to identify the predictors of improvement in patient skills or disease management, based on patient characteristics, IBD features, and treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with ulcerative colitis and Crohn's disease for more than 3 months, with a confirmed diagnosis according to European guidelines, being followed in the gastroenterology department at Saint Antoine Hospital.
* Aged over 18 years.
* Undergoing a multimodal day hospital visit, regardless of the scheduled intervention in the gastroenterology department at Saint Antoine Hospital.
* Not opposed to participating in the research.

Exclusion Criteria:

* Protective measure in place.
* Patient who has previously participated in an equivalent day hospital program.
* Pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ulcerative colitis and Crohn's disease for more than 3 months, with a confirmed diagnosis according to European guidelines, being followed in the gastroenterology department at Saint Antoine Hospital and eligible for a multimodal day hospital
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a change in their skills at one month or a modification in the management of their disease | 1 month
  For this study, the benefit of the multimodal Day Hospital (DH) will be evaluated through two groups of criteria:
  * The criteria of the "Improvement of Patient Skills" group, assessed at the time of day hospitalization and one month later.
  * The criteria of the "Improvement in Patient Management" group, assessed at the time of day hospitalization. The multimodal DH will be considered beneficial if at least one of these two groups of criteria is met.

SECONDARY OUTCOMES:
self-declared drug adherence rate | 1 and 6 month
  Evaluation of skill-related criteria at the 6-month mark self-declared drug adherence rate: scale from 0 to 100 A threshold below 80% defines non-compliant patients. A relative increase of 20% will be considered a significant improvement.
Percentage of patients requiring a treatment discontinuation | 1 and 6 month
Percentage of patients requiring changes in treatment dosages | 1 and 6 month
The proportion of patients showing improvement for each individual item. | 1 and 6 months
The total number of improved criteria per patient. | 1 and 6 months
The proportion of patients with access to practitioners such as a dietitian specialized in IBD, a rheumatologist, or a dermatologist, outside of the Day Hospital (DH) | 1 and 6 months
IBD-KID2 score | 1 and 6 month
  Understanding of disease and treatment based on the IBD-KID2 (inflammatory bowel disease knowledge inventory device) score, comprising 13 questions An absolute increase in score of 3 units will be considered a significant improvement
SLQF score for SLFQ Dietary Behavior Change | 1 and 6 month
  Patients are categorized into four knowledge categories: insufficient, problematic, sufficient, or excellent, based on respective scores of 0-25, 25-33, 33-42, and 42-50. Any move to a higher category will be considered a significant improvement.
Change in fatigue behaviors assessed using the Functional Assessment Chronic Illness Therapy-Fatigue (FACIT-F) | 1 and 6 month
  An absolute increase in score of 4 units will be considered a significant improvement
Work Productivity and Activity Impairment Questionnaire in Crohn's disease (WPAI:CD) | 1 and 6 month
  Change in work effectiveness behaviors assessed by the Work Productivity and Activity Impairment Questionnaire in Crohn's disease (WPAI:CD) An absolute increase in score of 20 units will be considered a significant improvement.
Work Productivity and Activity Impairment Questionnaire in in Ulcerative Colitis (WPAI:UC) | 1 and 6 month
  Change in work Productivity and Activity Impairment Questionnaire in Ulcerative Colitis (WPAI:UC) An absolute increase in score of 20 units will be considered a significant improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mclellan, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de gastroentérologie Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No
The questionnaires will be completed directly by the patients using an electronic platform accessible via the Internet (e-CRF Cleanweb - Telemedicine SA, with the "ePro" feature), developed by URCEST in collaboration with the coordinating investigator. This method of data collection was chosen to facilitate the completion process and streamline the questionnaire flow. A report of anonymized aggregated data at the end of the study will be published.
  No individual participant data will be available.